CLINICAL TRIAL: NCT04004546
Title: Improving Medication Adherence Through a Health Literacy-based Intervention for Coronary Heart Disease Patients With Low Health Literacy
Brief Title: Improving Medication Adherence Through a Health Literacy-based Intervention for Coronary Heart Disease Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: National Taiwan University (Other)
Responsible Party: Principal Investigator, Elaine Siow, Professional Consultant, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 4750368
Record Dates: First submitted 2019-06-27; First posted 2019-07-02 (Actual); Last update posted 2019-07-02 (Actual); Status verified 2019-06

CONDITIONS: Coronary Disease
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): At baseline: video and education booklet. 2-weeks after enrollment: telephone call by nurse.
  Interventions: Behavioral: Health literacy-based intervention
- Control group (No Intervention): Usual care

INTERVENTIONS:
Behavioral: Health literacy-based intervention — Participants in the intervention group will receive a: i) 30-min video about medication adherence, ii) medication adherence booklet, and iii) 2-week telephone call by a nurse.
  Arms: Intervention group

SUMMARY:
This is a multi-center pilot study to examine the effectiveness of a health literacy-based intervention to improve medication adherence and self-efficacy of medication use among individuals with coronary heart disease (CHD). The specific aims are to: i) develop a health literacy-based intervention to improve medication adherence for CHD individuals with low health literacy and ii) evaluate the effects of a health literacy-based intervention on improving medication adherence and self-efficacy in CHD individuals.

DETAILED DESCRIPTION:
The project will be conducted in 2 phases. Phase 1 is to develop the health literacy-based intervention that consists of a video and an education booklet. Phase 2 is to conduct a pilot study to evaluate the effectiveness of the intervention. A total of 60 participants with low health literacy and diagnosed with CHD will be recruited in two settings. Data will be collected at baseline and 4-weeks after enrollment. The following data will be collected:

At baseline: Socio-demographic information (e.g. age, gender, education level, income, past medical history, social support), health literacy (eligibility screening at time of recruitment), CHD knowledge, medication adherence, and medication self-efficacy.

4-weeks after enrollment: medication self-efficacy and medication adherence.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 years and diagnosed with CHD.
* Currently receiving pharmacological therapy such as statins, anti-platelet and/or blood thinner, beta-blockers, calcium channel blockers, nitroglycerin, and angiotensin- converting enzyme inhibitors (ACE).
* Low health literacy score of 9 or less as measured using the short-form Mandarin Health Literacy Scale (s-MHLS).

Exclusion Criteria:

* History of significant cognitive impairment, psychiatric disorders, and aphasia.
* Without access to a telephone or unable to give telephone contact.
* Currently enrolled in another program or clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-03-18 (Actual); Primary Completion 2019-09-30 (Estimated); Study Completion 2019-09-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline medication adherence at 4-weeks follow-up | Baseline and 4-weeks follow-up
  Measured using the Chinese version of the Hill-Bone Medication Adherence Scale (HB-MAS). The HB-MAS is a self-reported measure of the extent of medication adherence. The HB-MAS consists of 9 questions with each item rated on a 4-point scale (1 = none of the time; 2 = some of the time; 3 = most of the time; and 4 = all of the time). The total score ranges from 9 (minimum) to 36 (maximum), where lower scores indicate higher levels of medication adherence.

SECONDARY OUTCOMES:
Change from baseline medication self-efficacy at 4-weeks follow-up | Baseline and 4-weeks follow-up
  Measured using the Chinese version of the Self-Efficacy for Appropriate Medication Use (C-SEAMS). The C-SEAMS is a self-reported measure of the extent of confidence in taking medications. The C-SEAMS consists of 13 questions with each item rated on a 3-point scale (1 = not confident; 2 = somewhat confident; 3 = very confident). The total score ranges from 13 (minimum) to 39 (maximum), where higher scores indicate higher levels of self-efficacy for medication use.

OTHER OUTCOMES:
Health literacy | Baseline
  Measured using the short-form Mandarin Health Literacy Scale (s-MHLS). The s-MHLS consists of 11 questions to determine an individual's functional health literacy in terms of their ability to read, comprehend, and utilize basic health information in making personal health decisions. The sum of correct responses range from 0 (minimum) to 11 (maximum), where higher scores indicate higher levels of health literacy. Individuals with a total score of 9 or less are considered as having low health literacy.
Perceived social support | Baseline
  Measured using the Chinese version of the Medical Outcomes Study social support survey (MOS-SSS-C). The MOS-SSS-C consists of 19 items that measure 4 subscales of social support: emotional/informational support, tangible support, affectionate support, and positive social interaction. Participants are required to rate each item on a 5-point scale (1 = none of the time; 2 = a little of the time; 3 = some of the time; 4 = most of the time; 5 = all of the time). The average of the 4 subscale scores will be used to calculate the overall score that ranges from 0 (minimum) to 100 (maximum), where higher scores indicate better perceived social support.
CHD knowledge | Baseline
  Measured using the modified Chinese version of the knowledge inventory (m-CKI). The m-CKI is used to assess the individual's knowledge about CHD. The m-CKI consists of 32 multiple-choice questions with 5 options for each question. The sum of correct responses range from 0 (minimum) to 32 (maximum), where higher scores indicate better knowledge about CHD.

CONTACTS AND LOCATIONS:
Overall Officials: Elaine Siow, PhD, Principal Investigator — Chinese University of Hong Kong; Chang Nien-Tzu, PhD, Principal Investigator — National Taiwan University
Locations (2):
- The Nethersole School of Nursing, The Chinese University of Hong Kong, Shatin, New Territories, Hong Kong
- School of Nursing, National Taiwan University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No